CLINICAL TRIAL: NCT06994806
Title: A Phase 1, Open-label, Multicenter, Dose Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of KQB168 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Malignancies
Brief Title: A Study to Investigate the Safety and Efficacy of KQB168 as Monotherapy and in Combination in Participants With Advanced Solid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kumquat Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KQB168-101
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor Malignancies
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy Dose Escalation (Experimental): Drug: KQB168 - Oral KQB168
  Interventions: Drug: KQB168
- Combo Therapy Dose Escalation (Experimental): Drug: KQB168 - Oral KQB168 Drug: pembrolizumab - Intravenous pembrolizumab
  Interventions: Drug: KQB168; Drug: Pembrolizumab

INTERVENTIONS:
Drug: KQB168 — Oral KQB168
Drug: Pembrolizumab — Intravenous pembrolizumab
  Arms: Combo Therapy Dose Escalation

SUMMARY:
The goal of this clinical trial is to learn if KQB168 works to treat advanced solid tumor cancer in adults. It will also learn about the safety of KQB168. The main questions it aims to answer are:

* What is the safe dose of KQB168 by itself or in combination with pembrolizumab?
* Does KQB168 alone or in combination with pembrolizumab decrease the size of the tumor?
* What happens to KQB168 in the body?

Participants will:

* Take KQB168 daily, alone or in combination with pembrolizumab
* Visit the clinic about 8 times in the first 8 weeks, and then once every 3 weeks after that

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of solid tumor malignancy.
* Unresectable or metastatic disease that has progressed on immunotherapy.
* No available treatment with curative intent
* Adequate organ function
* Measurable disease per RECIST v1.1

Exclusion Criteria:

* Active primary central nervous system tumors
* Cardiac abnormalities
* History of lung diseases
* Any condition that may impair drug absorption or prevent oral dosing
* Known history of immune-mediated colitis and uncontrolled autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experience treatment-emergent adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) | up to 36 months
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of AEs, SAEs, and DLTs, from first dose of study treatment to 30 days after last dose of study treatment.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 36 months
  Using RECIST v1.1
Duration of response (DOR) | up to 36 months
  Using RECIST v1.1
Time to response (TTR) | up to 36 months
  Using RECIST v1.1
Disease control rate (DCR) | up to 36 months
  Using RECIST v1.1
Progression-free survival (PFS) | up to 36 months
  Using RECIST v1.1
Overall survival (OS) | up to 36 months
  using RECIST v1.1
Concentration-time curve (AUC) | up to 36 months
Maximum plasma concentration (Cmax) | up to 36 months
Time to maximum plasma concentration (tmax) | up to 36 months
Pharmacologically Active Dose (PAD) | up to 36 months
  Assessment of tumor and systemic immune activation

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - NEXT Austin, Austin, Texas
  - NEXT Huston, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No